CLINICAL TRIAL: NCT04882163
Title: A Phase 1B/2 Randomized, Multicenter, Open-Label Study Of Iberdomide (CC-220) In Combination With Polatuzumab Vedotin Plus Rituximab Or Tafasitamab Or Rituximab Plus Chemotherapy For Subjects With Relapsed Or Refractory Aggressive B-Cell Lymphoma
Brief Title: Study to Evaluate Tolerability of Iberdomide (CC-220) in Combination With Polatuzumab Vedotin Plus Rituximab or Tafasitamab or Rituximab Plus Chemotherapy in B-cell Lymphoma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business objectives have changed
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC-220-DLBCL-002; 2020-005333-32 (EudraCT Number)
Record Dates: First submitted 2021-05-06; First posted 2021-05-11 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Lymphoma, B-Cell
Keywords: CC-220; Phase 1B/2; B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — iberdomide; polatuzumab vedotin; Rituximab; tafasitamab; Gemcitabine; Cisplatin; Dexamethasone; Bendamustine Hydrochloride; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- CC-220 + Polatuzumab vedotin + rituximab- Cohort A (Experimental): Subjects with Relapsed or refractory (R/R) Aggressive B-cell lymphoma (a-BCL) will receive CC-220 at a dose specified by cohort dose level in combination with polatuzumab vedotin plus rituximab.
  Interventions: Drug: CC-220; Drug: Polatuzumab vedotin; Drug: Rituximab
- CC-220 + Tafasitamab- Cohort B (Experimental): Subjects with R/R a-BCL will receive CC-220 at a dose specified by cohort dose level in combination with tafasitamab.
  Interventions: Drug: CC-220; Drug: Tafasitamab
- CC-220 + Rituximab + Chemo (Cohort C) (Experimental): Subjects with R/R a-BCL will receive CC-220 at a dose specified by cohort dose level in combination with rituximab plus chemotherapy (Gemcitabine, cisplatin, dexamethasone).
  Interventions: Drug: CC-220; Drug: Rituximab; Drug: Gemcitabine; Drug: Cisplatin; Drug: Dexamethasone
- CC-220 + Pola + Ritux vs Pola + Benda + Ritux (Cohort D) (Experimental): Subjects will be randomized to receive either CC-220 + Pola (polatuzumab vedotin) + Ritux (rituximab) or polatuzumab vedotin + bendamustine + rituximab in 21-day treatment cycles. CC-220 will be given at the RP2D declared in Part 1 of this study. Polatuzumab vedotin and rituximab will be administered at the same levels as in part 1. Bendamustine will be given to subjects randomized in the control arm at a dose of 90 mg/m2 IV on Days 1 and 2 of each of the first 6 cycles.
  Interventions: Drug: CC-220; Drug: Polatuzumab vedotin; Drug: Rituximab; Drug: Bendamustine
- CC-220 + tafasitamab vs Lenalidomide + Tafasitamab- Cohort E (Experimental): Subjects will be randomized to receive either CC-220 + tafasitamab or lenalidomide + tafasitamab in 28-day treatment cycles. CC-220 will be given at the RP2D declared in Part 1 of this study and the tafasitamab will be at the same levels as in Part 1. Lenalidomide will be administered to subjects randomized in the control arm at a dose of 25 mg/day orally, for 21 days out of 28, for up to 12 cycles.
  Interventions: Drug: CC-220; Drug: Tafasitamab; Drug: Lenalidomide
- CC-220 + Rituximab + Chemo vs Rituximab + Chemo (Cohort F) (Experimental): Subjects will be randomized to receive either CC-220 + rituximab + chemotherapy (Gemcitabine, Cisplatin, Dexamethasone) or rituximab + chemotherapy (Gemcitabine, Cisplatin, Dexamethasone) in 21-day treatment cycles. CC-220 will be administered at the RP2D declared in Part 1 of this study and the combination medicines will be at the same levels as in part 1.
  Interventions: Drug: CC-220; Drug: Rituximab; Drug: Gemcitabine; Drug: Cisplatin; Drug: Dexamethasone

INTERVENTIONS:
Drug: CC-220 — CC-220
  Other Names: Iberdomide
Drug: Polatuzumab vedotin — Polatuzumab vedotin
  Arms: CC-220 + Pola + Ritux vs Pola + Benda + Ritux (Cohort D); CC-220 + Polatuzumab vedotin + rituximab- Cohort A
Drug: Rituximab — Rituximab
  Arms: CC-220 + Pola + Ritux vs Pola + Benda + Ritux (Cohort D); CC-220 + Polatuzumab vedotin + rituximab- Cohort A; CC-220 + Rituximab + Chemo (Cohort C); CC-220 + Rituximab + Chemo vs Rituximab + Chemo (Cohort F)
Drug: Tafasitamab — Tafasitamab
  Arms: CC-220 + Tafasitamab- Cohort B; CC-220 + tafasitamab vs Lenalidomide + Tafasitamab- Cohort E
Drug: Gemcitabine — Gemcitabine
  Arms: CC-220 + Rituximab + Chemo (Cohort C); CC-220 + Rituximab + Chemo vs Rituximab + Chemo (Cohort F)
Drug: Cisplatin — Cisplatin
  Arms: CC-220 + Rituximab + Chemo (Cohort C); CC-220 + Rituximab + Chemo vs Rituximab + Chemo (Cohort F)
Drug: Dexamethasone — Dexamethasone
  Arms: CC-220 + Rituximab + Chemo (Cohort C); CC-220 + Rituximab + Chemo vs Rituximab + Chemo (Cohort F)
Drug: Bendamustine — Bendamustine
  Arms: CC-220 + Pola + Ritux vs Pola + Benda + Ritux (Cohort D)
Drug: Lenalidomide — Lenalidomide
  Arms: CC-220 + tafasitamab vs Lenalidomide + Tafasitamab- Cohort E

SUMMARY:
This is a Phase 1b/2 randomized study of Iberdomide (CC-220) added to 3 different combination regimens (polatuzumab vedotin plus rituximab (Cohort A), tafasitamab (Cohort B), rituximab plus gemcitabine and platinum-based chemotherapy (Cohort C)) for participants with relapsed or refractory aggressive B-cell lymphoma (R/R a-BCL). All 3 cohorts will be open for enrollment at study start. Part 1 (dose escalation) will be followed by Part 2 (dose expansion), in which participants will be randomized to one of three cohorts, with CC-220 at the recommended Phase 2 Dose in combination with the Cohorts A, B and C treatment that is compared to their individual standard of care regimen.

ELIGIBILITY:
Inclusion Criteria:

* Participants must satisfy the following criteria to be enrolled in the study:

  1. Participant is ≥ 18 years of age at the time of signing the informed consent form (ICF).
  2. Participant has histologically confirmed (per local evaluation) diagnosis of, aggressive B-cell lymphoma (a-BCL) according to 2016 WHO classification among the following subtypes:

     1. Diffuse large B-cell lymphoma (DLBCL), Not otherwise specified (NOS) including Germinal center B-cell and Activated B-cell types;
     2. High-grade B-cell lymphoma, with MYC and B-cell lymphoma 2 (BCL2) and/or B-cell lymphoma 6 (BCL6) rearrangements;
     3. Primary mediastinal (thymic) large B-cell lymphoma (PMBCL);
     4. Primary cutaneous DLBCL-leg type;
     5. Anaplastic lymphoma kinase positive (ALK+) large B-cell lymphoma;
     6. Epstein Barr virus positive (EBV+) DLBCL, NOS;
     7. Grade 3b Follicular lymphoma (FL).
  3. Participants must have relapsed or refractory disease after at least 2 prior lines of therapy including Rituximab, cyclophosphamide, doxorubicin hydrochloride, vincristine sulfate, and prednisone (R-CHOP)-like regimen OR after one prior line of standard therapy and being not eligible for autologous stem cell transplant (ASCT); participants previously treated with CAR-T therapy can be enrolled.
  4. Participant must have measurable disease defined by at least one FDG-avid lesion for FDGavid-subtype and one bi-dimensionally measurable (> 1.5 cm in longest diameter) disease by computed tomography (CT) or magnetic resonance imaging (MRI), as defined by the Lugano classification (Cheson, 2014).
  5. Participant has an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
  6. Participant must have the following laboratory values:

     1. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L or ≥ 1.0 x 109/L in case of documented bone marrow involvement (> 50% or tumor cells), without growth factor support for 7 days (14 days if pegylated granulocyte-colony stimulating factor (peg-G-CSF))
     2. Hemoglobin ≥ 8 g/dL
     3. Platelets ≥ 75 x 109/L or ≥ 50 x 109/L in case of documented bone marrow involvement (> 50% or tumor cells), without transfusion for 7 days
     4. Aspartate aminotransferase / serum glutamic oxaloacetic transaminase (AST/SGOT) and alanine aminotransferase / serum glutamic pyruvic transaminase (ALT/SGPT) ≤ 2.5 x ULN except in the case of documented liver involvement by lymphoma, where ALT/SGPT and AST/SGOT must be ≤ 5.0 x ULN.
     5. Serum total bilirubin ≤ 2.0 mg/dL (34 μmol/L) except in cases of Gilbert syndrome, then ≤ 5.0 mg/dL (86 μmol/L)
     6. Estimated serum creatinine clearance of ≥ 50 mL/minute using the modification of diet in renal disease formula.
  7. All participants must:

     1. Have an understanding that the study drug could have a potential teratogenic risk.
     2. Agree to follow all requirements defined in the Pregnancy Prevention Program for CC-220 Pregnancy Prevention Plan for Participants in Clinical Trials.
  8. A female of childbearing potential (FCBP) must:

     a. Have two negative pregnancy tests as verified by the investigator prior to starting study therapy. She must agree to ongoing pregnancy testing during the course of the study, and after end of study therapy.
  9. Male participants must:

     1. Practice true abstinence (which must be reviewed on a monthly basis and source documented) or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study.

Exclusion Criteria:

* The presence of any of the following will exclude a participant from enrollment:

  1. Participant has any significant medical condition, active infection (including SARS-CoV-2 suspected or confirmed), laboratory abnormality, or psychiatric illness that would prevent the participant from participating in the study.

     a. In the case of prior SARS-CoV-2 infection, symptoms must have completely resolved
  2. Participant has any condition including the presence of laboratory abnormalities, which places the participant at unacceptable risk if he/she were to participate in the study.
  3. Participant has any other subtype of lymphoma.
  4. Participant has received systemic anti-cancer treatment, CAR-T or any T-cell targeting treatment (approved or investigational) ≤ 5 half-lives or 4 weeks prior to starting CC-220, whichever is shorter.
  5. Participant has received prior therapy with a Cereblon-modulating drug (eg, lenalidomide, avadomide) ≤ 4 weeks prior to starting CC-220.
  6. Participant has persistent diarrhea or malabsorption ≥ Grade 2 (NCI-CTCAE v5.0), despite medical management.
  7. Participant has peripheral neuropathy ≥ Grade 2 (NCI CTCAE v5.0).
  8. Participant is on chronic systemic immunosuppressive therapy or corticosteroids.
  9. Participant has impaired cardiac function or clinically significant cardiac disease.
  10. Participant had major surgery ≤ 2 weeks prior to starting CC-220.
  11. Participant has known seropositivity for or active viral infection with human immunodeficiency virus (HIV).
  12. Participant has known chronic active hepatitis B
  13. Participant has history of other malignancy, unless being free of the disease for ≥ 3 years prior to starting study drug; exceptions to the ≥ 3-year time limit include history of the following:

      1. Localized non-melanoma skin cancer
      2. Carcinoma in situ of the cervix
      3. Carcinoma in situ of the breast
      4. Incidental histologic finding of prostate cancer (T1a or T1b as per Tumor Node Metastasis [TNM] staging system) or prostate cancer that has been treated with curative intent.
  14. Participant has current treatment with strong CYP3A4/5 modulators.
  15. Participant has known hypersensitivity to any component of planned combination medications in the regimen.
  16. Participant has known allergy to thalidomide, pomalidomide, lenalidomide or avadomide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-10 (Estimated); Primary Completion 2026-04-08 (Estimated); Study Completion 2029-04-07 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | During the First cycle (each cycle is 28 days)
  Frequency of dose limiting toxicities (DLT) to define MTD of CC- 220 in combination with polatuzumab vedotin plus rituximab or tafasitamab or rituximab plus chemotherapy in subjects with R/R a-BCL.
Recommended Phase 2 Dose (RP2D) | During the First cycle (each cycle is 28 days)
  Frequency of dose limiting toxicities (DLT) to establish the RP2D of CC- 220 in combination with polatuzumab vedotin plus rituximab or tafasitamab or rituximab plus chemotherapy in subjects with R/R a-BCL.
Best Overall Response Rate (ORR) | Up to 7 years
  The proportion of participants with best overall response achieved during the study as either Complete Response or Partial Response before subsequent anti-lymphoma therapy.

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) | From enrollment until at least 28 days after last dose of study treatment
  An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a participant during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the participant's health, including laboratory test values regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a preexisting condition) should be considered an AE.
Best ORR- Part 1 | Up to 6 years
  The proportion of participants with best overall response achieved during the study as either Complete Response or Partial Response before subsequent anti-lymphoma therapy.
Complete Response Rate (CRR)- Part 2 | Up to 7 years
  The proportion of participants experiencing Complete Response before receiving any subsequent anti-lymphoma therapy.
Time to Response (TRR)- Part 2 | Up to 7 years
  The time from entry to the study (enrollment date for Part 1 and randomization date for Part 2) to the date of first documented response (≥ PR).
Duration of Response (DOR)- Part 2 | Up to 7 years
  The time from the earliest date of documented response (≥ PR) to the first occurrence of relapse or progression.
Progression-free Survival (PFS)- Part 2 | Up to 7 years
  The time from entry to the study (enrollment date for Part 1 and randomization date for Part 2) to the first occurrence of disease progression or death from any cause.
Overall Survival (OS)- Part 2 | Up to 7 years
  The time from entry to the study (enrollment date for Part 1 and randomization date for Part 2) to death from any cause.
Pharmacokinetics (PK) - Cmax | Up to 4 weeks
  Observed maximum CC-220 serum concentration
EORTC QLQ-C30 - Part 2 | Up to 7 years
  European Organization for Research and Treatment of Cancer - Quality of Life C30 questionnaire (EORTC QLQ-C30) consists of 30 questions incorporated into five functional domains (physical, role, cognitive, emotional, and social), nine symptom scales (fatigue, pain, nausea and vomiting, dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties), and a single global QoL/global health status score.
FACT-Lym LymS - Part 2 | Up to 7 years
  Functional Assessment of Cancer Therapy-Lymphoma Lymphoma subscale (FACT-Lym LymS) is a 15-item subscale that addresses health-related quality of life symptoms for Non-Hodgkin's lymphoma participants (eg, swelling, night sweats). The FACT instruments use a 5-point intensity type of rating scale (from "not at all" to "very much").
FACT/GOG-NTX-4 - Part 2 | Up to 7 years
  Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity 40-item questionnaire (FACT/GOG-NTX-4) is a 4-item peripheral neuropathy subscale used to differentiate between participants with and without treatment-related neurotoxicity. The FACT instruments use a 5-point intensity type of rating scale (from "not at all" to "very much").
EQ-5D-5L - Part 2 | Up to 7 years
  EQ-5D-5L has 2 components: a descriptive system and a visual analogue scale (VAS). The instrument's descriptive system consists of 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (27):
- United States (3):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Avera Cancer Institute, Sioux Falls, South Dakota
- Austria (2):
  - Medizinische Universität Graz, Graz
  - Universitätsklinikum St. Pölten, Sankt Pölten
- Belgium (3):
  - Cliniques Universitaires Saint-Luc, Brussels
  - Hôpital de Jolimont, La Louvière
  - H.-Hartziekenhuis Roeselare-Menen vzw, Roeselare
- France (5):
  - EDOG - Institut Bergonie - PPDS, Bordeaux
  - Hôpital François Mitterand, Dijon
  - Centre Hospitalier Lyon Sud, Lyon
  - EDOG - Institut Claudius Regaud - PPDS, Toulouse
  - Gustave Roussy, Villejuif
- South Korea (3):
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Seoul National University Hospital, Seoul
- Spain (4):
  - Hospital Universitario Germans Trias i Pujol, Badalona
  - Hospital Universitario 12 de Octubre, Madrid
  - Complejo Asistencial Universitario de Salamanca - H. Clinico, Salamanca
  - Hospital Universitario Virgen del Rocio - PPDS, Seville
- Taiwan (3):
  - Taipei Veterans General Hospital, Beitou District, Taipei City
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei, Zhongzheng Dist.
- United Kingdom (4):
  - Beatson West of Scotland Cancer Centre, Glasgow Scotland
  - Royal Liverpool University Hospital, Liverpool
  - Nottingham University Hospitals NHS Trust, Nottingham
  - University Hospital Southampton NHS Foundation Trust - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/